CLINICAL TRIAL: NCT05908903
Title: A Clinical Study on the Improvement of Sleep Quality, Skin Condition and Life Status After Taking Sleep Aid Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Botanee Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Botanee
Record Dates: First submitted 2023-05-29; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Sleep Disorder
Keywords: Sleep quality and skin conditions
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Skin Diseases | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Take drinks with active ingredients such as poria and GABA. Drink half an hour before bedtime, 10ml/bag/day, daily.
  Interventions: Combination Product: Drinks with active ingredients such as poria and GABA
- Control product group (Placebo Comparator): Take a control drink that does not contain GABA and poria. Drink half an hour before bedtime, 10ml/bag/day, daily.
  Interventions: Combination Product: Drinks with active ingredients such as poria and GABA

INTERVENTIONS:
Combination Product: Drinks with active ingredients such as poria and GABA — Take drinks half an hour before bedtime, 10ml/bag/day, daily. Subjects are uniformly using skin care products provided by the sponsor during the test.

SUMMARY:
The main objective of the study is to observe changes in the subjects' sleep quality, skin condition and life status after 4 weeks of using a sleep aid drink (AOXMED Poria γ-aminobutyric acid drink).

This is a single-center, randomized, double-blind, controlled, 4-week (28-day) clinical study conducted in Chinese healthy women aged 25-55 years old who were offered a sleep aid drink.

DETAILED DESCRIPTION:
The study population is 70 healthy Chinese women aged 25-55 years with a PSQI ≥ 7 (presence of sleep disorder) who report current problems with dryness, roughness, dullness and lack of elasticity on their face. The subjects will be randomly divided into an experimental group and a control product group of 35 subjects each, and the distribution of age and total hours of sleep will be more or less equal in both groups.

Subjects will be formally enrolled after on-site assessment and will undergo follow-up site visits and test product administration. During the test cycle, subjects in the experimental group will take a drink with the active ingredients of Poria, Poria and GABA, and subjects in the control product group will take a control drink without Poria, Date Palm and GABA ingredients for 4 weeks. To avoid the influence of different skincare products on the results, all subjects will be asked to use the basic skincare products with only moisturizing ingredients provided by the sponsor during the test period. The efficacy of the test products will be verified by comparing the changes in sleep quality, skin condition and life status of the subjects before and after taking the test products for 2 and 4 weeks, and by comparing the differences in sleep quality, skin condition and life status between the test and control groups.

ELIGIBILITY:
Inclusion Criteria:

1. 25-55 years old, Chinese female;
2. PSQI index ≥ 7 (presence of sleep disorders);
3. The subject's self-reported facial problems such as dryness, roughness, dullness, and lack of elasticity;
4. The BMI of the subjects was between 18~24kg/m2;
5. After the doctor's clinical evaluation, there are mild facial skin roughness (1 point and above) and mild to moderate overall facial wrinkles (3~6 points);
6. Corneometer base measurement of facial skin moisture in 15~45 (Corneometer Unit, C.U.) Between;
7. Have basic Chinese reading ability;
8. can use smartphones;
9. Be in good health and free of any other chronic diseases other than skin problems and sleep disorders or diseases being treated;
10. Voluntarily participate in the test and sign the informed consent form; 11） Willingness to comply with all evaluation requirements;

Exclusion Criteria:

1. Products with anti-wrinkle, firming, repairing and nourishing effects are not included in the skin care products used;
2. Intend to become pregnant, or are pregnant or breastfeeding;
3. Have a history of alcoholism;
4. Have a history of allergies;
5. Participated in any clinical trial evaluation within 1 month;
6. Those who have applied any anti-inflammatory drugs to the test site within the past two months;
7. Those who have suffered from skin diseases (such as psoriasis, eczema, psoriasis, skin cancer, etc.);
8. patients with insulin-dependent diabetes;
9. Patients with asthma or other chronic respiratory diseases who are being treated;
10. Have taken/injected anti-allergic drugs in the past 1 month;
11. Patients who have received anti-cancer chemotherapy or immunotherapy patients within the past 6 months;
12. Have any other health problems or chronic diseases;
13. Applying retinoids, A hydroxy acids, salicylic acids, hydroquinone within the past 3 months, or prescription drugs (antibiotics, retinoids, A hydroxy acids and steroids) in use within the past 6 months, oral contraceptives (if you have been taking the same contraceptive pills for the past 6 months, you can continue to take them);
14. Experts or professionals believe that there are other iatrogenic reasons that will affect the evaluation results; 15) Those who have undergone surgery, plastic surgery or organ transplantation in the past year.

Ages: 25 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Identification by Chinese ID card
Enrollment: 70 (Actual)
Dates: Start 2022-07-09 (Actual); Primary Completion 2022-08-07 (Actual); Study Completion 2022-08-07 (Actual)

PRIMARY OUTCOMES:
Changes in the Pittsburgh Sleep Quality Index | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline PSQI index at 2 weeks by questionnaire. Obtain change from Baseline PSQI index at 4 weeks by questionnaire.
Changes in the sleep duration | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline sleep duration at 2 weeks by sleep quality monitoring bracelet.
  Obtain change from Baseline sleep duration at 4 weeks by sleep quality monitoring bracelet.
Sleep Quality Assessment after 2-week application | Week2
  Obtain data on agreement with sleep improvement by sleep quality self-assessment questionnaire
Sleep Quality Assessment after 4-week application | Week4
  Obtain data on agreement with sleep improvement by sleep quality self-assessment questionnaire

SECONDARY OUTCOMES:
Changes in the skin hydration | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline skin hydration at 2 weeks by Corneometer. Obtain change from Baseline skin hydration at 4 weeks by Corneometer.
Changes in the skin glossiness | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline skin glossiness at 2 weeks by Glossymeter. Obtain change from Baseline skin glossiness at 4 weeks by Glossymeter.
Changes in the skin firmness | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline skin firmness at 2 weeks by cutometer. Obtain change from Baseline skin firmness at 4 weeks by cutometer.
Changes in the skin elasticity | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline skin elasticity at 2 weeks by cutometer. Obtain change from Baseline skin elasticity at 4 weeks by cutometer.
Changes in the individual type angle | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline Individual type angle at 2 weeks by Colorimeter. Obtain change from Baseline Individual type angle at 4 weeks by Colorimeter.
Changes in the proportion of crow's feet area | Week0（Baseline）、Week2、Week4
  Calculate the proportion of crow's feet area by Visia CR images. Obtain change from Baseline proportion of crow's feet area at 2 weeks. Obtain change from Baseline proportion of crow's feet area at 4 weeks.
Changes in the proportion of fine lines under the eye | Week0（Baseline）、Week2、Week4
  Calculate the proportion of fine lines under the eye by Visia CR images. Obtain change from Baseline proportion of fine lines under the eye at 2 weeks. Obtain change from Baseline proportion of fine lines under the eye at 4 weeks.
Changes in the degree of wrinkle severity | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline degree of wrinkle severity at 2 weeks by Dermatologist evaluation according to Skin Aging ATLAS of Asian Type.
  Obtain change from Baseline degree of wrinkle severity at 4 weeks by Dermatologist evaluation according to Skin Aging ATLAS of Asian Type.
Changes in the grade of skin dryness | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline grade of skin dryness at 2 weeks by Dermatologist evaluation according to 5-point dryness scale.
  Obtain change from Baseline grade of skin dryness at 4 weeks by Dermatologist evaluation according to 5-point dryness scale.
Changes in the CIE RGB of skin tone | Week0（Baseline）、Week2、Week4
  Dermatologist use PANTONE SkinTone (Pantone color card) skin color guide to evaluate skin tone grade of subjects. Find the CIE RGB corresponding to the skin tone grade in Pantone ColorManager software and convert it into a color value using the formula for data analysis: CIE RGB = R+G*256+B*256*256.
  Calculate the change from Baseline CIE RGB of skin tone at 2 weeks. Calculate the change from Baseline CIE RGB of skin tone at 4 weeks.
Skin condition Assessment after 2-week application | Week2
  Obtain data on agreement with skin condition improvement by skin condition self-assessment questionnaire
Skin condition Assessment after 4-week application | Week4
  Obtain data on agreement with skin condition improvement by skin condition self-assessment questionnaire
Changes in the satisfaction with the quality of life | Week0（Baseline）、Week2、Week4
  Obtain change from Baseline satisfaction with the quality of life at 2 weeks accessed by WHOQOL-100 questionnaire.
  Obtain change from Baseline satisfaction with the quality of life at 4 weeks accessed by WHOQOL-100 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Song Weiming, Master, Principal Investigator — Yan Shu Medical Beauty Chain Group
Locations (1):
- Shanghai China-norm Quality Technical Service Co ，Ltd, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Data is used to develop new products, no decision has been made on when to disclose